CLINICAL TRIAL: NCT02111525
Title: Fluid Status of Outpatients With Dyspnea
Acronym: FLOOD
Status: Completed | Type: Observational
Sponsor: Intersection Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-000030
Record Dates: First submitted 2014-04-08; First posted 2014-04-11 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Dyspnea,; Acute Heart Failure Syndrome; Pulmonary Congestion
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the distribution of lung fluid status as reported by the IMED-4 system in patients presenting to the emergency department or urgent care facility with shortness of breath.

ELIGIBILITY:
INCLUSION CRITERIA

* Shortness of breath as the most prominent presenting symptom
* Age greater ≥ 45
* Willingness, ability, and commitment to participate in the study

EXCLUSION CRITERIA

* Patients with any active implantable medical device
* Patients who are pregnant or lactating
* Patients who have tattoos and or non-intact skin directly under the electrode position
* Patients who have had past allergic reactions to medical grade adhesives
* Patients that are dialysis dependent
* Patients who have had a lung lobectomy
* Patients in whom the shortness of breath presentation is due to obvious non HF cause such as acute chest trauma
* Patients who have received nitrates (sub-lingual, topical or IV), diuretics or vasopressors ≥ 1 hour prior to IMED-4 Recording
* Patients who decline to have their backs photographed with the IMED-4 device in position
* Patients who are receiving invasive or non-invasive positive airway pressure (PAP) ventilation prior to or following presentation to the ED (Self presentation or admission via EMS).
* Severe co-morbidity or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, incarceration, shortened life expectancy, etc.)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with shortness of breath to an emergency department or urgent care facility are possible candidates for the study and shall be screened for suitability based on the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Lung Fluid Status | Up to 1 year
  The IMED 4 is a new device designed to measure the lung fluid status by assessing how wet or dry the lungs are

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wayne State University Hospital, Detroit, Michigan
  - Vanderbilt University, Nashville, Tennessee